CLINICAL TRIAL: NCT00726856
Title: A Retrospective Survey to Evaluate the Effectiveness and Safety of Dual Inhibition Lipid-lowering Regimen in the Treatment of Dyslipidemic Patients in Normal Practice
Brief Title: Retrospective Survey Evaluating the Effectiveness and Safety of Dual Inhibition Lipid-lowering in the Treatment of Dyslipidemia (Study P05171)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P05171
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Ezetimibe; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Fenofibrate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: patients with dyslipidemia
  Interventions: Drug: Ezetimibe 10 mg plus statin or ezetimibe 10 mg plus fenofibrate

INTERVENTIONS:
Drug: Ezetimibe 10 mg plus statin or ezetimibe 10 mg plus fenofibrate — Ezetimibe 10 mg taken daily for 3 months
  Other Names: SCH 58235

SUMMARY:
This retrospective study evaluates the effectiveness and safety of ezetimibe plus statin or ezetimibe plus fenofibrate in dyslipidemic patients that were treated with these dual inhibition lipid lowering regimens as part of their normal standard of care. This study assesses the percentage of patients who achieve LDL-C target goals and also evaluates the patient compliance to treatment.

DETAILED DESCRIPTION:
Retrospective medical chart review

ELIGIBILITY:
Inclusion Criteria:

* Patient was > 20 years and < 75 years of age on the index date*
* Patient diagnosed with dyslipidemia who did not respond adequately based on NCEP ATP III target to previous lipid lowering treatment, and have received dual inhibition therapy, such as ezetimibe plus statins, ezetimibe plus fenofibrate or ezetimibe alone, for at least 3 months
* Patient has at least one Total Cholesterol and LDL-C measurements at baseline and 3 months after initiating the dual inhibition therapy.
* Patient has the following records documented in the chart during the data collection period:

  * Medical history and co morbidities (if available)
  * Total Cholesterol and LDL-C. test results before and after initiating the dual inhibition therapy
  * Prescription information of lipid-lowering dual inhibition regimens NOTE: * Index date: the date of initiating dual inhibition therapy

Exclusion Criteria:

* Patients who do not meet all the inclusion criteria will be excluded from this survey.
* Patients who were enrolled in other clinical trial observing specific study procedures which deviates from normal practice will not be included in this study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with dyslipidemia who did not respond adequately based on NCEP ATP III target to previous lipid lowering treatment, and have received dual inhibition therapy, such as ezetimibe plus statins, ezetimibe plus fenofibrate or ezetimibe alone, for at least 3 months
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2007-05; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the change in LDL-C levels after treatment | 3 months

SECONDARY OUTCOMES:
Assessment of the percentage of patients who attain their National Cholesterol Education Program (NCEP) Adult Treatment Panel (ATP) III target for LDL-C | 3 months
Assessment of patient compliance by evaluating the length of stay on therapy | 3 months
Comparison of the patient comorbidities among populations gathered from different levels of hospitals and specialties | 3 months
Evaluation of safety and tolerability in patients receiving dual inhibition therapy | 3 months